CLINICAL TRIAL: NCT00885287
Title: Study of Therapeutic Efficacy, Safety and Pharmacokinetic Interactions Between Artemether-lumefantrine and Nevirapine-based Antiretrovirals in HIV-infected Patients With Uncomplicated Falciparum-malaria in Muheza, Northeastern Tanzania
Brief Title: Interactions Between Artemether-lumefantrine and Antiretrovirals in HIV-patients With Uncomplicated Malaria in Tanzania
Acronym: InterACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Lasse Vestergaard, Dr, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIMR/HQ/R.8a/Vol.IX/794
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Malaria, Falciparum; HIV Infections
Keywords: uncomplicated malaria; HIV/AIDS; drug interactions; antimalarial drug efficacy; antiretrovirals; pharmacovigilance; Tanzania
MeSH Terms: conditions — Malaria, Falciparum; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HIV-positives on ARVs receiving AL for malaria (Active Comparator): HIV-positive patients on first-line ARVs receiving artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria
  Interventions: Drug: Artemether-lumefantrine (AL)
- HIV-positives receiving AL for malaria (Active Comparator): HIV-positive patients not receiving antiretrovirals but receiving artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria
  Interventions: Drug: Artemether-lumefantrine (AL)
- HIV-negatives receiving AL for malaria (Active Comparator): HIV-negative patients receiving artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria
  Interventions: Drug: Artemether-lumefantrine (AL)

INTERVENTIONS:
Drug: Artemether-lumefantrine (AL) — Standard treatment-dose of artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria according to national treatment guidelines

SUMMARY:
As HIV/AIDS is spreading in malaria-endemic countries, many patients here will need concomitant treatment for both infections. Effective combination treatments are available for both malaria (artemisinin-based combination treatments, ACTs) and HIV/AIDS (antiretroviral combination treatments, ARTs), and these treatments are presently recommended for concomitant use by ministries of health in many endemic countries, including Tanzania. However, theoretically some of these drugs may be involved in harmful interactions with each other, as they share common cytochrome enzymes involved in their metabolism. Such interactions could lead to less effective treatments and/or adverse effects, as a consequence of reduced or increased drug levels, respectively. Only little clinical and pharmacological information is however yet available to guide clinicians and policy-makers on this issue.

The main aim of the InterACT study in Tanzania is to conduct a series of detailed observational studies of clinical and paraclinical safety, therapeutic efficacy and pharmacokinetic interactions between the currently nationally recommended first-line treatment for malaria, artemether-lumefantrine, and first-line antiretroviral treatments, primarily nevirapine-based combinations, for HIV/AIDS. The studies will be conducted among patients with uncomplicated malaria, who attend the HIV/AIDS Care and Treatment Clinic and Muheza Designated District Hospital in Muheza, north-eastern Tanzania, which is an area characterized by intense transmission of Plasmodium falciparum malaria and with a prevalence of HIV around 8-10%. The study is expected to inform guidelines for the treatment of malaria in patients with HIV/AIDS in Tanzania, and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive and HIV-negative patients with confirmed P. falciparum infection in the presence of either measured fever (> 37.5°C) or a history of fever within the previous 24 hours; for HIV-positive patients also afebrile patients are eligible in the presence of other symptoms of malaria (e.g., coughing, diarrhea, headache, nausea, body weakness, body pain).
* Not being pregnant or lactating.
* Absence of history of clinically significant hypersensitivity reactions to any of the study medicines being evaluated.
* For HIV-positive patients on cART, successful adherence to treatment without prominent adverse events for a period of a minimum of six weeks prior to the date of enrollment will be required.
* Easy access to the health facility (travel time < 1 hour) and the ability to attend the stipulated follow-up visits.
* Informed consent provided by the patient or by a parent/guardian

Exclusion Criteria:

* Patients below body weight of 10 kilograms (for under fives).
* Existence of underlying chronic severe illness (e.g., cardiac, renal or hepatic disease).
* No use within the previous four weeks prior to enrollment of any other antimalarial or other drug with antimalarial activity (with the exception of drugs required as part of standard treatment of HIV/AIDS, e.g., sulfamethoxazole and trimethoprim).

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 830 (Actual)
Dates: Start 2009-07; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Clinical and parasitological efficacy of artemether-lumefantrine; incidence and severity of treatment-related clinical and paraclinical adverse events; changes in pharmacokinetic profiles of artemether-lumefantrine. | 42 days of post-treatment follow-up

SECONDARY OUTCOMES:
Changes in pharmacokinetic profiles of nevirapine-based and other used antiretrovirals; | 42 days of post-treatment follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Vestergaard, MD, PhD, Principal Investigator — University of Copenhagen; Martha Lemnge, PhD, Principal Investigator — National Institute for Medical Research, Tanzania
Locations (1):
- Muheza Designated District Hospital, Muheza, Tanga, Tanzania